CLINICAL TRIAL: NCT03060382
Title: The Treatment of Knee Osteoarthritis With Balanced Buttress Absorbable Spacer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DP2017
Record Dates: First submitted 2017-02-18; First posted 2017-02-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-02

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- balanced buttress absorbable spacer (Experimental): For the patients of study group, a balanced buttress absorbable spacer was placed into tibia.
  Interventions: Device: balanced buttress absorbable spacer
- total knee arthroplasty (Placebo Comparator): For the patients of control group, total knee arthroplasty was conducted.
  Interventions: Biological: total knee arthroplasty

INTERVENTIONS:
Device: balanced buttress absorbable spacer — For the patients of study group, a balanced buttress absorbable spacer was placed into the gap after the osteotomy of tibia and fibula to modify the lower limb line.
  Arms: balanced buttress absorbable spacer
Biological: total knee arthroplasty — Total knee arthroplasty was conducted for the patients of control group
  Arms: total knee arthroplasty

SUMMARY:
The investigators randomly divided the knee osteoarthritis patients met the inclusive criteria into two groups (study group and control group). Placement of balanced buttress absorbable spacer and total knee arthroplasty were conducted. The clinical outcome of two groups were compared in this study.

DETAILED DESCRIPTION:
Knee osteoarthritis, caused by non-uniform settlement of medial and lateral tibial plateau, was not uncommon in clinic. Medial stenosis was the most type of the disease. The symptoms included knee pain during walking and varus deformity of lower limbs. Total knee arthroplasty and tibial osteotomy were two common conventional treatment of the knee osteoarthritis, which were not minimally invasive and bring great financial burden to patients' family. The investigators planned to recruit 150 patients of knee osteoarthritis into this study, which were randomly divided into two groups (study group and control group). For the patients of study group, a balanced buttress absorbable spacer was placed into the gap after the osteotomy of tibia and fibula to modify the lower limb line. However, total knee arthroplasty was conducted for the patients of control group. The patients were followed up and the clinical outcomes were compared in this study.

ELIGIBILITY:
Inclusion Criteria:

* 40-80 years old
* Medial stenosis of the knee
* Varus deformity less than 20 degrees

Exclusion Criteria:

* Lateral stenosis of the knee
* Hepatic renal dysfunction
* Refuse to participate the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
functional outcome | 12 months
  walking distance the patients could bear

SECONDARY OUTCOMES:
complication | 1 week
  vascular nerve bundle injury

CONTACTS AND LOCATIONS:
Overall Officials: Yingze Zhang, M.D, Study Chair — Third Hospital of Hebei Medical University Department of Orthopaedic Surgery; Zhiyong Hou, M.D, Study Director — Third Hospital of Hebei Medical University Department of Orthopaedic Surgery; Ruipeng Zhang, M.D, Principal Investigator — Third Hospital of Hebei Medical University Department of Orthopaedic Surgery
Locations (2):
- China (2):
  - Hebei Medical University Third Hospital, Shijiazhuang, Hebei
  - Zhiyong Hou, Shijiazhuang, Hebei

IPD SHARING:
Plan to Share IPD: Yes